CLINICAL TRIAL: NCT05203939
Title: A Phase 1/2 Study to Assess the Safety and Efficacy of OCU400 for Retinitis Pigmentosa Associated With NR2E3 and RHO Mutations and Leber Congenital Amaurosis With Mutation(s) in CEP290 Gene
Brief Title: Study to Assess the Safety and Efficacy of OCU400 for Retinitis Pigmentosa and Leber Congenital Amaurosis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OCU400-101
Record Dates: First submitted 2021-11-16; First posted 2022-01-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Retinitis Pigmentosa; Leber Congenital Amaurosis
Keywords: NR2E3; Rhodopsin; Enhanced S-cone syndrome; Cep290
MeSH Terms: conditions — Retinitis Pigmentosa; Leber Congenital Amaurosis; Night Blindness, Congenital Stationary, Autosomal Dominant 1; Enhanced S-Cone Syndrome; Meckel Syndrome, Type 4

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Low Dose) (Experimental): Biallelic autosomal recessive NR2E3 mutations subgroup or Autosomal dominant NR2E3 mutation or RHO mutations subgroup
  Interventions: Drug: OCU400 Low Dose
- Cohort 2 (Mid Dose) (Experimental): Biallelic autosomal recessive NR2E3 mutations subgroup or Autosomal dominant NR2E3 mutation or RHO mutations subgroup
  Interventions: Drug: OCU400 Med Dose
- Cohort 3 (High Dose) (Experimental): Biallelic autosomal recessive NR2E3 mutations subgroup or Autosomal dominant NR2E3 mutation, RHO mutations subgroup
  Interventions: Drug: OCU400 High Dose
- Pediatric Arm (Experimental): Pediatric subjects will receive the medium dose concentration
  Interventions: Drug: OCU400 Med Dose
- Phase 2 (High and Medium Dose) (Experimental): Following DSMB confirmation, adult RP subjects with Biallelic autosomal recessive NR2E3 mutations, autosomal dominant NR2E3 mutations, Autosomal dominant RHO mutations will receive a high dose concentration of OCU400 or LCA patients with CEP290 mutation will receive a medium dose concentration of OCU400.
  Interventions: Drug: OCU400 Med Dose; Drug: OCU400 High Dose
- Adult Arm (Experimental): Biallelic autosomal recessive NR2E3 mutations subgroup or Autosomal dominant NR2E3 mutation, RHO mutations subgroup will receive a high dose concentration of OCU400 and LCA patients with CEP290 will receive a medium dose concentration of OCU400
  Interventions: Drug: OCU400 Med Dose; Drug: OCU400 High Dose
- Second Eye Dosing (Experimental): Eligible RP participants will be dosed in the untreated fellow eye with a therapeutic dose used in Phase 3 study of OCU400 (1.0x10E11vg/mL in 250 μl ) and will be followed for an additional 48 weeks.
  Interventions: Drug: OCU400 Second Eye Dosing
- Natural History Study (OCU400-104) (No Intervention): A Prospective and Retrospective Natural History Study of RP and LCA:
  This is an observatory study for the prospective natural history of RP and LCA in adult and pediatric subjects. The study will also collect and review retrospective data and ophthalmology examination of natural history and progression of disease for all subjects starting with earliest timepoint on or after the date of their diagnosis of RP or LCA.
  Subjects will be seen up to a total of four times during the 12 months of the Observational Period, at baseline, 3 months, 6 months and 12 months.
  A total of up to 100 subjects will be enrolled in the study, including:
  Approximately 76 newly enrolled subjects consisting of 50 adult RP subjects, 6 adult LCA subjects, 20 pediatric RP/LCA subjects. Up to 24 subjects that reconsent from the OCU400-101 study (subjects from OCU400-101 will provide data on their untreated eye)

INTERVENTIONS:
Drug: OCU400 Low Dose — subretinal injection of up to 1.66×10E10 vg/mL
  Arms: Cohort 1 (Low Dose)
Drug: OCU400 Med Dose — subretinal injection of up to 3.33×10E10 vg/mL
  Arms: Adult Arm; Cohort 2 (Mid Dose); Pediatric Arm; Phase 2 (High and Medium Dose)
Drug: OCU400 High Dose — subretinal injection of up to 1.66×10E11 vg/mL
  Arms: Adult Arm; Cohort 3 (High Dose); Phase 2 (High and Medium Dose)
Drug: OCU400 Second Eye Dosing — subretinal injection of 1.0x10E11vg/mL in 250 μl
  Arms: Second Eye Dosing

SUMMARY:
This is a Phase 1/2 Study to Assess the Safety and Efficacy of OCU400 in patients with retinitis pigmentosa associated with NR2E3 and RHO mutations and in patients with LCA due to mutation(s) in CEP290 gene (OCU400-101). To document prospective eye pathology in the above subjects Investigators will also conduct a Natural History Study (OCU400-104)i

This is a multicenter study, which will be conducted in two phases and will enroll up to a total of 24 subjects in the OCU400-101 and 100 subjects in the OCU400-104 study.

DETAILED DESCRIPTION:
This study will be conducted in two phases enrolling up to 24 subjects. Treated subjects will receive a single subretinal injection of OCU400 in the study eye.

This is a multicenter, open-label, dose-ranging study in two subgroups of subjects with three consecutive cohorts.

A total of 18 adult RP subjects from each of the following subgroups with Biallelic autosomal recessive NR2E3 mutations, autosomal dominant NR2E3 mutations or Autosomal dominant RHO mutations will be selected for dose escalation.

For the Phase I portion of the study, the 3+3 design for sequential dose-escalating cohorts will be used with scheduled 3 dosing levels between 9 and 18 subjects will be used to follow the design.

Up to 3 additional adult LCA patients with CEP290 mutations and at least 1 pediatric LCA subject, will be enrolled in the Phase 2 portion.

Sample Size Justification:

The trial will enroll up to 24 patients (18 adult RP, up to 3 LCA patients, and at least 1 pediatric LCA patient) in both Phase 1 and Phase 2 components.

Participants who meet eligibility criteria will be enrolled and receive a single subretinal injection of OCU400 in one study eye. Participants are considered to have completed this study if they complete the final EOS visit Week 48 (12 months following the IP dose). The study duration will be approximately 58 weeks for each participant and will be followed in Long Term Safety Follow Up for an additional 2 years.

Participants from the Phase 1/2 study who previously received the investigational product (OCU400) in one eye may be eligible to receive OCU400 in the untreated fellow eye, provided they meet the inclusion/exclusion criteria and have completed week 48 follow up visit.

Natural History Study (OCU400-104, A Prospective and Retrospective Natural History Study of RP and LCA):

This is an observatory study for the prospective natural history of RP and LCA in adult and pediatric subjects. The study will also collect and review retrospective data and ophthalmology examination of natural history and progression of disease for all subjects starting with the earliest timepoint on or after the date of their diagnosis of RP or LCA. Enrollment for this study has closed.

ELIGIBILITY:
Diagnosis and main criteria for inclusion:

Subjects meeting all inclusion criteria and none of the exclusion criteria are eligible for study participation.

Inclusion Criteria for Adult RP:

1. Males or females ≥ 18 years of age at the time of informed consent.
2. Confirmed genetic diagnosis of biallelic autosomal recessive NR2E3 mutations or autosomal dominant NR2E3 mutation for Subgroup 1 or autosomal dominant RHO mutations for Subgroup 2.
3. For the sentinel subject of Cohort 1-3, BCVA ≤ 20/160 in study eye or visual field less than 20° in any meridian, as measured by a III4e isopter or equivalent in study eye.
4. For non-sentinel subject, BCVA ≤ 20/50 or visual field less than 20° in any meridian, as measured by a III4e isopter or equivalent in study eye.
5. Able to perform a Multi-Luminance Mobility Testing (MLMT) using study eye, but unable to pass the MLMT at 1 lux, the lowest luminance level tested.

Exclusion Criteria for Adult RP:

1. Subject lacks evidence of outer nuclear layer.
2. Considered unsuitable for any reason that may either place the subject at increased risk during participation or interfere with the interpretation of the study outcomes by the Investigator, or the Sponsor after reviewing medical, ocular, and psychiatric history, clinical examination, and laboratory evaluation, as determined by the Investigator.
3. Previous treatment with a gene therapy or cell therapy product.
4. Previous treatment with any investigational drug or device within one year.
5. Any contraindications for subretinal injection.
6. Cataract Surgery within 3 months. YAG capsulotomy within 1 month. Any other intraocular surgery within 6 months.
7. Breast-feeding, pregnancy, sperm donation or inability to practice strict contraception within the Treatment Observation Period.
8. Any medical condition with life expectancy < 6 years.

Inclusion Criteria for Adult LCA:

1. Males or females at least 18 years of age at the time of informed consent.
2. Clinical diagnosis of LCA and confirmed genetic diagnosis of CEP290 mutation.
3. Best corrected visual acuity (BCVA) equal to or worse than LogMAR +0.7 but equal to or better than LogMAR 3.8 (light perception) in the study eye.
4. Detectable outer nuclear layer in the macular region as determined by spectral-domain optical coherence tomography (SD-OCT).

Exclusion Criteria for Adult LCA:

1. Any symptom of central nervous system involvement/disease that would impact the ability to measure visual function.
2. Considered unsuitable for any reason that may either place the patient at increased risk during participation or interfere with the interpretation of the study safety and efficacy outcomes by the Investigator, after reviewing medical, ocular, and psychiatric history, clinical examination, and laboratory evaluation, as determined by the Investigator.
3. Any contraindications for subretinal injection.
4. Any intraocular surgery within 6 months.
5. Active ocular/intraocular infection (e.g., conjunctivitis, keratitis, scleritis, endophthalmitis).
6. Breast-feeding, pregnancy, sperm donation or inability to practice strict contraception within the Treatment Observation Period.

Inclusion Criteria for Pediatric RP:

1. Males or females 6 - 17 years of age (inclusive) at the time of parental permission and/or assent, whichever is applicable.
2. Confirmed genetic diagnosis of biallelic autosomal recessive NR2E3 mutations or autosomal dominant NR2E3 mutation for Subgroup 1 or autosomal dominant RHO mutations for Subgroup 2.
3. BCVA ≤ 20/32 or visual field less than 20° in any meridian, as measured by a III4e isopter or equivalent in study eye.
4. Able to perform a Multi-Luminance Mobility Testing (MLMT) using study eye, but unable to pass the MLMT at 1 lux, the lowest luminance level tested.

Exclusion Criteria for Pediatric RP:

1. Subject lacks evidence of outer nuclear layer as determined by spectral-domain optical coherence tomography (SD-OCT).
2. Considered unsuitable for any reason that may either place the subject at increased risk during participation or interfere with the interpretation of the study outcomes by the Investigator, or the Sponsor after reviewing medical, ocular, and psychiatric history, clinical examination, and laboratory evaluation, as determined by the Investigator.
3. Previous treatment with a gene therapy or cell therapy product.
4. Previous treatment with any investigational drug or device within one year.
5. Any contraindications for subretinal injection.
6. Cataract surgery within 3 months. YAG capsulotomy within 1 month. Any other intraocular surgery within 6 months.
7. Breast-feeding, pregnancy, or inability to practice strict contraception within the Treatment Observation Period for subjects of childbearing potential.
8. Active ocular/intraocular infection (e.g., conjunctivitis, keratitis, scleritis, endophthalmitis).
9. Any medical condition with life expectancy < 6 years.

Inclusion Criteria for Pediatric LCA:

1. Males or females 6 - 17 years of age (inclusive) at the time of parental permission and/or assent, whichever is applicable.
2. Clinical diagnosis of LCA and confirmed genetic diagnosis of CEP290 mutation.
3. Best corrected visual acuity (BCVA) equal to or worse than LogMAR +0.7 but equal to or better than LogMAR 3.8 (light perception) in the study eye.
4. Detectable outer nuclear layer in the macular region as determined by spectral-domain optical coherence tomography (SD-OCT).

Exclusion Criteria for Pediatric LCA:

1. Any symptom of central nervous system involvement/disease that would impact the ability to measure visual function.
2. Considered unsuitable for any reason that may either place the subject at increased risk during participation or interfere with the interpretation of the study safety and efficacy outcomes by the Investigator, after reviewing medical, ocular, and psychiatric history, clinical examination, and laboratory evaluation, as determined by the Investigator.
3. Any contraindications for subretinal injection.
4. Any Intraocular surgery within 6 months.
5. Active ocular/intraocular infection (e.g., conjunctivitis, keratitis, scleritis, endophthalmitis).
6. Breast-feeding, pregnancy, or inability to practice strict contraception within the Treatment Observation Period for subjects of childbearing potential.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Study Drug-related adverse events (SDAE) | 1 year
  Counts, frequencies and percentages of SDAEs. SDAE is a primary adverse event of interest and defined as AEs and SAEs that are direct subjects to the Study Drug only.
Treatment-Emergent adverse events (TEAEs) | 1 year
  Counts, frequencies and percentages TEAEs. TEAEs are defined as an event that was not present prior to administration of the dose of study drug and present after the dose, or if it represents the exacerbation of an event that was present prior to the dose.
Serious adverse events (SAEs) | 1 year
  Counts, frequencies and percentages of SAEs including Resulted in Death, Life-threatening, Hospitalization, Disabling/incapacitating, Congenital anomaly or birth defect and medically significant AEs ( AE that did not meet any of the above criteria but could have jeopardized the subject and might have required medical or surgical intervention to prevent one of the outcomes listed above).

SECONDARY OUTCOMES:
Best-corrected visual acuity (BCVA) | 1 year (Changes from baseline)
  Measured as the ETDRS letter score on the EVA tester or E-ETDRS charts. Electronic ETDRS Visual Acuity Testing Protocol will be followed (confidential).
Low-luminance visual acuity (LLVA) | 1 year (Changes from baseline)
  Electronic Visual Acuity Tester (EVA) and a Sponsor specific Low-Luminance lens will be used. Early Treatment of Diabetic Retinopathy Study (ETDRS) will also be accepted as a backup.
Slit-lamp biomicroscopy | 1 year (Changes from baseline)
  Changes in visual function.
Intraocular pressure (IOP) | 1 year (Changes from baseline)
  IOP measurement by applanation or rebound tonometry. Confirmation with Goldmann tonometer if IOP reading is outside the normal range (8-21mmHg).
Indirect ophthalmoscopy | 1 year (Changes from baseline)
  If visual acuity is so poor that the participant is unable to count fingers or perceive hand motion, light perception will be tested with the indirect ophthalmoscope as the light source.
anti-AAV5 (anti Adeno-associated virus type 5) | 1 year
  Blood samples will be collected for the assessment. These samples will be analyzed using validated assays at a bioanalytical laboratory.
anti-hNR2E3 antibodies (hNR2E3 gene) | 1 year
  Blood samples will be collected for the assessment. These samples will be analyzed using validated assays at a bioanalytical laboratory.
T-cell response | 1 year
  Blood samples will be collected for the assessment. These samples will be analyzed using validated assays at a bioanalytical laboratory.

OTHER OUTCOMES:
Multi-luminance mobility testing (MLMT) | 1 year (Changes from baseline)
  Subjects will navigate a standardized mobility maze under set conditions as specified times during the study. The mobility testing will follow a standardized administration and data acquisition protocol and may only be administered by site staff certified in the methodology.
Changes in ellipsoid zone width/length on wide-field 20° SD-OCT | 1 year (Changes from baseline)
  Ellipsoid zone area/outer segment length will be determined by Spectral Domain Optical Coherence Tomography (SD-OCT) using standardized systems and acquisition protocols.
Contrast sensitivity | 1 year (Changes from baseline)
  Contrast sensitivity will be conducted using Pelli-Robson chart.
Full Field Light Stimulation Threshold (FST) | 1 year (Changes from baseline)
  FST will be completed at scheduled times throughout the study period
Photopic Static Visual Fields | 1 year (Changes from baseline)
  The Octopus 900 will be used with a standardized white-on-white full field and a blue-on-yellow with full field
Vision on Quality of Life | 1 year (Changes from baseline)
  The National Eye Institute Visual Function Questionnaire 25 (NEI-VFQ25) and the Michigan Retinal Degeneration Questionnaire (MRDQ) questionnaires (for RP Adult subjects only) will be administered to assess the impact of vision on quality of subject's life.
Full Field Electroretinogram | 1 year (Changes from baseline)
  The International Society for Clinical Electrophysiology of Vision (ISCEV) guidelines will be followed for conducting ff-ERG (Full-field Electroretinography) for RP subjects only.
Wide-field fundus autofluorescence (wf-FAF) | 1 year (Changes from baseline)
  The intensity of FAF will be evaluated using 55° posterior pole scanning.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Qamar, MD, MPH, CMI, Study Chair — Ocugen
Locations (7):
- United States (7):
  - Associated Retina Consultants, Phoenix, Arizona
  - Ocugen Site 5 - University of California, San Diego (UCSD) - Shiley Eye Institute, La Jolla, California
  - Ocugen Site 3 - Bascom Palmer Eye Institute, Miami, Florida
  - Ocugen Site 6 - Emory University, Atlanta, Georgia
  - Ocugen Site 2 - Casey Eye Institute - OHSU, Portland, Oregon
  - Ocugen Site 8 - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Ocugen Site 1 - Retina Foundation of the Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Retina World Congress 2024- Meeting Abstract. Title: Safety and Efficacy Results from a Phase 1/2 Clinical Trial of OCU400 Modifier Gene Therapy for Treatment of Retinitis Pigmentosa — https://ocugen.com/wp-content/uploads/2024/06/Poster-OCU400.pdf
- See also: ARVO Annual Meeting 2024- Meeting Abstract: Title: OCU400 Nuclear Hormone Receptor-Based Gene Modifier Therapy: Safety and Efficacy from Phase 1/2 Clinical Trial for Retinitis Pigmentosa Associated with NR2E3 and RHO Mutations — http://iovs.arvojournals.org/article.aspx?articleid=2796216
- See also: International Conference on Ophthalmology and Vision Science, Canada- Meeting Abstract: Title: Evaluation of Safety and Efficacy of OCU400 Gene Therapy for Retinitis Pigmentosa: Phase 1/2 Study Results — https://www.scitechseries.com/ophthalmology/uploads/pdfs/final-scientific-program.pdf
- See also: American Academy of Ophthalmology (AAO) Annual Meeting- Title: Safety and Efficacy of OCU400 Gene Modifier Therapy for Retinitis Pigmentosa: Phase 1/2 Study Updates — https://aao.apprisor.org/apsSession.cfm?id=PD15